CLINICAL TRIAL: NCT02005887
Title: A Randomized Phase II Trial Evaluating the Endocrine Activity and Efficacy of Neoadjuvant Degarelix Versus Triptorelin in Premenopausal Patients Receiving Letrozole for Primary Endocrine Responsive Breast Cancer
Brief Title: TRial on the Endocrine Activity of Neoadjuvant Degarelix
Acronym: TREND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 41-13; 2012-005326-29 (EudraCT Number)
Record Dates: First submitted 2013-11-08; First posted 2013-12-09 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer Invasive Nos
Keywords: Premenopausal patients; ER-positive; PgR+ (>50%); HER2-negative or not amplified
MeSH Terms: interventions — Triptorelin Pamoate; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triptorelin + letrozole (Experimental): Arm A: Triptorelin 3.75 mg i.m. on day 1 every 28 days for 6 cycles + letrozole 2.5 mg/day orally for 6 cycles
  Interventions: Drug: triptorelin; Drug: letrozole
- degarelix + letrozole (Experimental): Arm B: Degarelix 240 mg s.c. on day 1 of cycle 1, followed by 80 mg s.c. on day 1 of cycles 2 to 6 + letrozole 2.5 mg every day orally for 6 cycles
  Interventions: Drug: degarelix; Drug: letrozole

INTERVENTIONS:
Drug: triptorelin — Triptorelin 3.75 mg injected into the muscle on day 1 every 28 days for 6 cycles (1 cycle= 28 days)
  Other Names: decapeptyl
  Arms: triptorelin + letrozole
Drug: degarelix — Degarelix 240 mg injected under the skin given as two injections of 120 mg on the first day of treatment, followed by injection of 80 mg on day 1 of cycles 2 to 6 (1 cycle=28 days)
  Other Names: firmagon
  Arms: degarelix + letrozole
Drug: letrozole — Letrozole 2.5 mg orally every day for 6 cycles
  Other Names: femara

SUMMARY:
The purpose of the this study is to investigate the anti-tumor activity and tolerability of the study medications Degarelix and Triptorelin in premenopausal women receiving preoperative treatment with Letrozole.

DETAILED DESCRIPTION:
RATIONALE Preoperative chemotherapy enables breast-conserving surgery for some patients with breast cancer, and it might be advantageous in several other ways. For example, the response to primary treatment may be used as a prognostic marker, since it has been demonstrated to be associated with a longer disease-free survival (DFS) compared with no response. In particular the degree of response (pathological complete remission (pCR)) predicts overall outcome in terms of DFS.

However, pCR can be achieved only in a minority of patients with estrogen receptor (ER)-positive disease. Studies in the medical literature indicate that pCR rates range from 2% to 10% in those patients whose tumors express ER suggesting that objective response and decrease of Ki67 must be considered within this subset of tumors.

The results of phase II studies and randomized phase III trials have clearly shown that preoperative endocrine therapy is a feasible and safe option among patients with hormone-receptor positive tumors. Letrozole has been shown to induce greater rates of clinical responses and of breast-conserving surgery in postmenopausal women as compared with tamoxifen.

In premenopausal women with ER and progesterone receptor (PgR) positive breast cancer, the preoperative endocrine therapy includes a combination of a gonadotropin-releasing hormone analogue (GnRH) plus tamoxifen. Recent studies suggest that neoadjuvant endocrine therapy with a combination of GnRH analogue and aromatase inhibitors (AIs: letrozole or anastrozole) is effective in selected premenopausal patients. The GnRH analogue, also known as a luteinizing hormone-releasing hormone agonist (LHRH agonist) or LHRH analogue, is a synthetic peptide drug modeled after the human hypothalamic gonadotropin-releasing hormone (GnRH). A GnRH analogue is designed to interact with the GnRH receptor and modify the release of pituitary gonadotropins, follicle-stimulating hormone (FSH) and luteinizing hormone (LH) for therapeutic purposes. Upon administration of a GnRH analogue, an initial stimulating action of the hypophysis occurs - termed a "flare" effect - which eventually causes a paradoxical and sustained drop in gonadotropin secretion. This second effect has been termed "downregulation" and can be observed after about 10 days. While this phase is reversible following cessation of medication, it can be maintained when GnRH agonists' use is continued for a long time. For a select group of patients, there is a delay of approximately 2-4 months before downregulation of the gonadotropins is observed.

Degarelix (INN) or degarelix acetate (USAN) (tradename: Firmagon) is a hormonal therapy approved for the treatment of prostate cancer. Since testosterone, a male hormone, promotes the growth of many prostate tumors, reduction of circulating testosterone to very low (castration) levels is often the treatment goal in the management of advanced prostate cancer. Degarelix, an antagonist of GnRH, has immediate onset of action through binding to GnRH receptors in the pituitary gland and blocking their interaction with GnRH. The result is a fast and profound reduction in LH, FSH and in turn, testosterone suppression. Its activity in suppressing the ovaries of premenopausal women might therefore be faster than other GnRH analogues, possibly by several weeks. The probable difference in onset of action could have significant clinical value for patients who are candidates for short-term neoadjuvant endocrine treatment.

TRANSLATIONAL RESEARCH A tumor block from the diagnostic core biopsy and one from final surgery will be collected and banked for central review and future translational research at the IBCSG Tissue Bank hosted by the European Institute of Oncology in Milan, Italy.

PATIENT-REPORTED SYMPTOMS The patient-reported symptoms (PRS) will be assessed using the Functional Assessment of Cancer Therapy Endocrine Subscale (FACT-ES) comprising 18 items (each has score range from 0 to 4) with a possible maximum total score of 72. Functional Assessment of Chronic Illness Therapy (FACIT) guidelines will be used for scoring and interpretation of the FACT-ES total score. Patients will be asked to complete a PRS Form at baseline (prior to randomization), at day 1 of cycle 2, at day 1 of cycle 4, and prior to surgery.

The objectives are

* To assess the differences in PRS score over time between the two treatment arms
* To correlate the estradiol (E2) levels and total PRS score measured on day 1 of cycle 2 and day 1 of cycle 4 of triptorelin or degarelix administration
* To summarize each of the 18 individual (endocrine symptom) items of the FACT-ES descriptively over time as the proportion of patients with "clinically significant" symptoms (those scoring 3 or 4)

STRATIFICATION Stratification will be performed according to:

- Age(in years): less than or equal to 39 versus 40 or more

STATISTICAL CONSIDERATIONS To achieve the primary objective, E2 levels will be determined centrally from samples taken at day 1 of the first treatment cycle before the administration of the first dose of degarelix or triptorelin (baseline), and thereafter at 24 and 72 hours, 7 days and 14 days after the first injection, and on day 1 of cycles 2 to 6 before the administration of degarelix or triptorelin.

For sample size calculation, we assume that the cumulative percentages of patients in the triptorelin arm achieving optimal ovarian function suppression (defined as E2 ≤2.72 pg/mL or ≤10 pmol/L) will be 30% within 2 weeks, 60% within 4 weeks and 75% within 8 weeks, and that degarelix will provide more rapid suppression (i.e., 60% within 2 weeks, 95% within 4 weeks and 100% within 8 weeks). Enrollment of 25 patients in each treatment arm will provide at least 90% power to detect a difference in time to optimal ovarian function suppression between the two groups, using a two sample log-rank test with a two-sided significance level of 0.05.

Randomized patients who receive at least one injection of triptorelin or degarelix will be included in the primary analysis. The primary endpoint will be compared between the two treatment arms using a stratified two-sample log-rank test, with age as stratification factor. The distribution of the primary endpoint will be summarized using the method of Kaplan-Meier and the two-sided 95% confidence interval (CI) for the difference in proportion of patients who achieve optimal ovarian function suppression between the two treatment arms at the end of the 1st, 2nd and 4th cycle will also be provided.

The toxicity, changes in Ki67 expression levels, the Preoperative Endocrine Prognostic Index (PEPI) score at the time of surgery, disease response, node-negative disease status at surgery and breast-conserving surgery (BCS) rate will also be summarized and differences assessed between treatment arms with confidence intervals.

The primary endpoint for patient-reported symptoms (PRS) analysis is the total PRS score measured at baseline, day 1 of cycle 2 and day 1 of cycle 4 of triptorelin or degarelix administration, and prior to surgery. The differences in PRS measurements between the two treatment arms over time will be explored using the repeated measures analysis based on generalized estimating equation (GEE) model.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Premenopausal status measured within 14 days Prior to randomization: Estradiol (E2) must be above 54 pg/mL (or above 198 pmol/L
* Age ≥ 18 years
* Performance Status - Eastern Cooperative Oncology Group (ECOG) 0-1
* Histologically confirmed invasive breast cancer: Primary tumor greater than 2 cm Diameter, any nodal stage, no evidence of metastasis (M0)
* Primary tumor must have ER and PgR >50% of the cells
* Primary tumor must be HER2-negative (by IHC and/or ISH)
* Hematopoietic status: Absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, hemoglobin ≥ 9 g/dL
* Hepatic status: Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), AST and ALT ≤ 2.5 × ULN, Alkaline phosphatase ≤ 2.5 × ULN
* Renal status: Creatinine ≤ 1.5 ×ULN
* Negative serum pregnancy test, within 2 weeks (preferably 7 days) prior to randomization.
* The patient must be willing to use effective non-hormonal contraception after the pregnancy test and up to surgery. Oral, injectable, or implant hormonal contraceptives or medicated IUD are not allowed within 2 months prior to randomization and during the trial.
* Prior fertility treatment is allowed but must have been stopped at least 12 months before randomization.
* The patient has completed the baseline patient-reported symptoms questionnaire.
* Written Informed Consent (IC) must be signed and dated by the patient and the Investigator prior to randomization.
* The patient has been informed of and agrees to data transfer and handling, in accordance with national data protection guidelines.
* The patient accepts blood samples to be taken for the determination of the primary endpoint.
* The patient agrees to make tumor available for submission for central pathology review and for translational studies as part of this protocol

Exclusion Criteria:

* Postmenopausal
* Any hormonal treatment (e.g., oral, injectable, implant, or medicated IUD) in the previous 2 months
* Presence of HER2 overexpression or amplification
* Received any prior treatment for primary invasive breast cancer
* Received any GnRH analog or SERM or AI within 12 months prior to randomization
* A history of malignant neoplasms within the past 10 years, except for curatively treated,Basal and squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the bladder
* Previous ipsilateral breast cancer (invasive or in situ) at any time
* Inflammatory breast cancer
* Bilateral invasive breast cancer
* Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension (≥ 180/110), unstable diabetes mellitus, dyspnea at rest, or chronic therapy with oxygen
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety
* Unresolved or unstable, serious adverse events from prior administration of another investigational drug
* Active or uncontrolled infection CTCAE v.4 grade 2 or higher
* Dementia, altered mental status, or any psychiatric condition that would prevent the understanding or rendering of Informed Consent
* Treatment with an investigational agent must have stopped at least 30 days before randomization.
* Pregnant or lactating women; lactation has to stop before randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Dellapasqua, MD, Study Chair — European Institute of Oncology,Milan,Italy; Marco Colleoni, MD, Study Chair — European Institute of Oncology, Milan, Italy
Locations (7):
- Italy (7):
  - Azienda Ospedaliero-Universitaria Policlinico S. Orsola-Malpighi di Bologna, Bologna
  - Ospedali Galliera, Genova
  - Istituto Europeo di Oncologia, IEO, Milan
  - Salvatore Maugeri Fondation, Pavia
  - Istituto Toscana Tumori, Prato
  - Ospedale degli Infermi, Rimini
  - A.O "Ospedale di Circolo e Fondazione" Macchi, Varese

REFERENCES:
- [Background] Kaufmann M, von Minckwitz G, Mamounas EP, Cameron D, Carey LA, Cristofanilli M, Denkert C, Eiermann W, Gnant M, Harris JR, Karn T, Liedtke C, Mauri D, Rouzier R, Ruckhaeberle E, Semiglazov V, Symmans WF, Tutt A, Pusztai L. Recommendations from an international consensus conference on the current status and future of neoadjuvant systemic therapy in primary breast cancer. Ann Surg Oncol. 2012 May;19(5):1508-16. doi: 10.1245/s10434-011-2108-2. Epub 2011 Dec 23. PMID 22193884
- [Background] Fisher B, Bryant J, Wolmark N, Mamounas E, Brown A, Fisher ER, Wickerham DL, Begovic M, DeCillis A, Robidoux A, Margolese RG, Cruz AB Jr, Hoehn JL, Lees AW, Dimitrov NV, Bear HD. Effect of preoperative chemotherapy on the outcome of women with operable breast cancer. J Clin Oncol. 1998 Aug;16(8):2672-85. doi: 10.1200/JCO.1998.16.8.2672. PMID 9704717
- [Background] Guarneri V, Broglio K, Kau SW, Cristofanilli M, Buzdar AU, Valero V, Buchholz T, Meric F, Middleton L, Hortobagyi GN, Gonzalez-Angulo AM. Prognostic value of pathologic complete response after primary chemotherapy in relation to hormone receptor status and other factors. J Clin Oncol. 2006 Mar 1;24(7):1037-44. doi: 10.1200/JCO.2005.02.6914. PMID 16505422
- [Background] Kuerer HM, Newman LA, Smith TL, Ames FC, Hunt KK, Dhingra K, Theriault RL, Singh G, Binkley SM, Sneige N, Buchholz TA, Ross MI, McNeese MD, Buzdar AU, Hortobagyi GN, Singletary SE. Clinical course of breast cancer patients with complete pathologic primary tumor and axillary lymph node response to doxorubicin-based neoadjuvant chemotherapy. J Clin Oncol. 1999 Feb;17(2):460-9. doi: 10.1200/JCO.1999.17.2.460. PMID 10080586
- [Derived] Dellapasqua S, Gray KP, Munzone E, Rubino D, Gianni L, Johansson H, Viale G, Ribi K, Bernhard J, Kammler R, Maibach R, Rabaglio-Poretti M, Ruepp B, Di Leo A, Coates AS, Gelber RD, Regan MM, Goldhirsch A, Colleoni M; International Breast Cancer Study Group. Neoadjuvant Degarelix Versus Triptorelin in Premenopausal Patients Who Receive Letrozole for Locally Advanced Endocrine-Responsive Breast Cancer: A Randomized Phase II Trial. J Clin Oncol. 2019 Feb 10;37(5):386-395. doi: 10.1200/JCO.18.00296. Epub 2018 Dec 27. PMID 30589600

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Triptorelin + Letrozol: Arm A: Triptorelin 3.75 mg i.m. on day 1 every 28 days for 6 cycles + letrozole 2.5 mg/day orally for 6 cycles
  Triptorelin: Triptorelin 3.75 mg injected into the muscle on day 1 every 28 days for 6 cycles (1 cycle= 28 days)
  Letrozole: Letrozole 2.5 mg orally every day for 6 cycles
- Arm B: Degarelix + Letrozol: Arm B: Degarelix 240 mg s.c. on day 1 of cycle 1, followed by 80 mg s.c. on day 1 of cycles 2 to 6 + letrozole 2.5 mg every day orally for 6 cycles
  Degarelix: Degarelix 240 mg injected under the skin given as two injections of 120 mg on the first day of treatment, followed by injection of 80 mg on day 1 of cycles 2 to 6 (1 cycle=28 days)
  Letrozole: Letrozole 2.5 mg orally every day for 6 cycles
Period: Overall Study
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
Started | 26 | 25
Completed | 26 | 23
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44.0 [42.2 to 47.5] | 45.0 [42.0 to 50.0] | 44.0 [42.0 to 48.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Time to Optimal Ovarian Function Suppression
Description: Time from the first injection of degarelix or triptorelin to the first assessment of centrally assessed 17-β-estradiol (E2) level in the range of optimal ovarian function suppression (≤2.72 pg/mL or ≤10 pmol/L) during the 6 cycles of neoadjuvant treatments.
Time Frame: up to 24 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
Number analyzed (Participants) | 26 | 25
days | 14 [8 to 14] | 3 [3 to 3]

2. Secondary Outcome: Ki67 Proliferation Marker Changes
Description: The percent change in Ki67 expression from pre-treatment diagnostic (baseline) biopsy to surgery, calculated as (surgery-baseline)/baseline*100.
Time Frame: Before day1 of cycle 1 and surgery
Population: Four patients are not evaluable: two patients did not undergo surgery during trial period, two patients did not have specimen submitted from surgery
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
Number analyzed (Participants) | 25 | 22
percentage change | -10.0 [-15.0 to -5.0] | -8.0 [-15.8 to -4.2]

3. Secondary Outcome: Preoperative Endocrine Prognostic Index (PEPI) Score
Description: Preoperative Endocrine Prognostic Index (PEPI) is the sum of the risk points (tumor size, nodal status, Ki67 level, ER status) with a 0-12 score representing the best prognostic feature (0 being the best score; 12 being the worst score), as previously determined to be associated with recurrence-free survival.
Time Frame: After 24 weeks or the time of surgery
Population: Two patients who did not have surgery were not evaluated
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
Number analyzed (Participants) | 26 | 23
scores on a scale | 6.5 [4.0 to 7.0] | 6.0 [4.0 to 7.0]

4. Secondary Outcome: Best Overall (Disease) Response
Description: Based on WHO tumor measurement and response criteria [1], measured from the start of treatment across all time points until disease progression or the end of 6 cycles of neoadjuvant therapies, whichever comes first. Response was determined by the IBCSG Head of Medical Affairs. An internal review (IR) form was created to record the final determination on best overall response. Confirmation of partial or complete response by an additional scan was not required in this trial. Best overall response was assessed based on changes in tumor size from baseline to the assessments after 3 and after 6 cycles (denoted as day 1 of cycle 4 and prior to surgery respectively) as measured physically by caliper or ruler and as measured by breast tumor imaging (i.e., bilateral mammography and breast ultrasound).
Time Frame: From day 1 of cycle 1 across all time points until disease progression
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
Number analyzed (Participants) | 26 | 25
percentage of patients | 46.2 [30.1 to 62.2] | 44.0 [27.7 to 60.3]

5. Secondary Outcome: Percentage of Patients With Node-negative Disease at Surgery
Description: The number of lymph nodes assessed at surgery minus the number of positives nodes identified, equal to zero.
Time Frame: During surgery, an average of 2 hours
Population: Two patients who did not have surgery were not evaluated
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
Number analyzed (Participants) | 26 | 23
percentage of patients | 34.6 [19.3 to 50.0] | 43.5 [26.5 to 60.5]

6. Secondary Outcome: Percentage of Patients Who Underwent Breast-Conserving Surgery (BCS)
Description: Whether or not patient undergoes BCS (per Surgery form).
Time Frame: During surgery, an average of 2 hours
Population: Two patients who did not have surgery were not evaluated
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
Number analyzed (Participants) | 26 | 23
percentage of patients | 42.3 [26.4 to 58.2] | 52.2 [35.0 to 69.3]

7. Secondary Outcome: Patient-reported Symptoms (PRS) Outcomes
Description: The patient-reported symptoms (PRS) will be assessed using the Functional Assessment of Cancer Therapy Endocrine Subscale (FACT-ES) comprising 18 items (each has score range from 0 to 4) with a possible minimum total score of 0 and maximum total score of 72 (72 is best). Functional Assessment of Chronic Illness Therapy (FACIT) guidelines will be used for scoring and interpretation of the FACT-ES total score.
Time Frame: At baseline, day 1 of cycle 2 and cycle 4 and prior to surgery; cycle 4 reported
Population: All patients who received at least one dose of trial treatment and had at least one FACT-ES assessment were included in the analysis
Measure: Number (90% Confidence Interval); unit: units on a scale
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
Number analyzed (Participants) | 26 | 25
units on a scale | 64 [62 to 67] | 62 [59 to 64]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) forms were submitted at the end of every cycle (28 days) and 30 days after surgery. All patients submitted AE data during 6 cycles of treatment period when available.
Description: Adverse events were collected using CTCAE v4.0. Each targeted AE will be classified according to the maximum grade of the event while on trial treatment (grade 0,1,2,3,4,5; where 0=no report). Other grade 3-5 AEs will be classified according to the maximum grade of any reported other AE.
Arm/Group | Arm A: Triptorelin + Letrozol | Arm B: Degarelix + Letrozol
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 23/26 | 23/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Triptorelin + Letrozol (N=26) | Arm B: Degarelix + Letrozol (N=25)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 3 (3) | 1 (1)
Injection Site Reaction (General disorders) | 0 (0) | 6 (7)
Alanine Aminotransferase (ALT) (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 8 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (4) | 6 (6)
Vaginal Dryness (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Hot Flashes/Flushes (Vascular disorders) | 18 (18) | 20 (23)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT02005887/SAP_000.pdf
  • Study Protocol (2012-12-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT02005887/Prot_001.pdf